CLINICAL TRIAL: NCT04932863
Title: A Prospective Observational Non Interventional Study of Reactogenicity and Safety of the BNT162b2 Messenger Ribonucleic Acid (mRNA) Covid-19 Vaccine in Cancer Patients on Active Treatment
Brief Title: BNT162b2 Messenger Ribonucleic Acid (mRNA) Covid-19 Vaccine in Cancer Patients on Active Treatment
Acronym: UNICO
Status: Completed | Type: Observational
Sponsor: Ente Ospedaliero Ospedali Galliera (Other)
Collaborators: Universita degli Studi di Genova (Other)
Responsible Party: Principal Investigator, Andrea DeCensi, Director of Medical Oncology, Ente Ospedaliero Ospedali Galliera
Other Study IDs: 35UCS2021
Record Dates: First submitted 2021-06-14; First posted 2021-06-21 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Neoplasms; Cancer, Treatment-Related
Keywords: neoplasms; COVID-19; Pfizer SARS- CoV-2 RNA vaccine
MeSH Terms: conditions — Neoplasms; Neoplasms, Second Primary; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Lymphocytes B and T cells for antigen-specific immune response studies; serum for cytokine panel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects with cancer of any type and stage under active or prior medical treatment: BNT162b2 mRNA Covid-19 Vaccine as two injections, 21 days apart, of 30 μg per dose in the deltoid muscle.
  Interventions: Biological: BNT162b2 mRNA Covid-19 Vaccine

INTERVENTIONS:
Biological: BNT162b2 mRNA Covid-19 Vaccine — Two injections, 21 days apart, of the BNT162b2 vaccine 30 μg per dose in the deltoid muscle.

SUMMARY:
In this Italian observational study the antibody titer reactogenicity to Pfizer Severe Acute Respiratory Syndrome (SARS) - Coronavirus (CoV-2) RNA vaccine in cancer patients under active antitumor treatment will be evaluated at 21 and 42 days and after 6 months. Furthermore patients safety will be monitored. Factors affecting immunogenicity (or lack of), including cancer treatment, will be the primary aim of the study.

DETAILED DESCRIPTION:
This is an observational non-interventional study in cancer patients. The study will evaluate the safety, tolerability and immunogenicity of Pfizer SARS-CoV-2 RNA vaccine against COronaVIrus Disease-19 (COVID-19) which will be delivered in the deltoid muscle in 2-dose (separated by 21 days). Blood will be collected in two 5 milliliters (mL) vacuettes for serum Immunoglobulin G (IgG) and Cytokine assessment, at baseline and after 21 days, immediately before the first and the second dose, respectively, then after 42 days from the first dose and finally after 6 months from the baseline. A panel of 22 cytokines (Biorad) will be measured at baseline and after 21 and 42 days in four groups consisting of: no responders (S1/S2 IgG<15 Arbitrary Unit AU/ml at 42 days), slow responders (S1/S2 IgG<15 AU/mL after 21 days and >15 AU/mL after the second dose), fast responders (S1/S2 IgG>15 AU/mL after the first 21 days) and immunized patients (S1/S2 IgG>15 AU/mL at baseline). At baseline, at 42 days and 6 months questionnaires for psychological testing will be dispensed for completion to patients.

After 42 days from the first dose, 15 mL of heparinized peripheral blood from both non-responders (S1/S2 IgG<25 AU/mL) and responders will be used for isolation of different Cluster of Differentiation 4 (CD4+) and CD8+ T cell subpopulations and analysis of their capability to undergo activation/proliferation in response to specific SARS- CoV-2 derived peptides.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* On treatment for cancer during the last 6 months or being treated >6 months ago but being ultravulnerable
* About to receive "Pfizer-BioNTech COVID-19" vaccine
* Lymphocyte count≥0.5x10^9/L

Exclusion Criteria:

* Subjects who are not eligible for "Pfizer-BioNTech COVID-19" vaccine administration
* Inability and/or unwillingness to sign written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients on current or prior active treatment or ultravulnerable according to clinical characteristics
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Antibody titer reactogenicity assessment | up to 12 months
  Serum IgG assessment at baseline, after 21 days, 42 days and after 6 months to Pfizer SARS- CoV-2 RNA vaccine in cancer patients under prior or current active antitumor treatment
Comparison of the immune response in treated and untreated patients | up to 12 months
  Identification of predictive factors for antibody response in treated versus untreated patients

SECONDARY OUTCOMES:
Safety assessment | up to 24 months
  Number and Grade of Adverse Events (AE) related to vaccine in patients undergoing anti-cancer treatment.
Antibody titer correlations with therapy | up to 24 months
  To correlate the antibody titer with type and timing of therapy. Particular attention will be devoted to the effect in patients receiving checkpoint inhibitor immunotherapy.
Antibody titer correlations with cancer | up to 24 months
  To correlate the antibody titer with the type of cancer and cancer staging/grading
Antibody titer correlations with patients | up to 24 months
  To correlate the antibody titer with host characteristics, including psychological variables such as distress and anxiety or depression.
Inflammatory response evaluation | up to 24 months
  Dosage of soluble factors (including pro-inflammatory cytokines, Cytokine Multiplex Assay Kits) in responders and non responders to Pfizer SARS-CoV-2 RNA vaccine
Immune cell activation | up to 24 months
  Correlate soluble factors of inflammatory response with blood cell count and inflammatory and pro-thrombotic biomarkers
Immunological memory | up to 24 months
  Comparing lymphocyte activation in cancer patients responding to the vaccine versus those non responding (S1/S2 IgG <15 AU/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea De Censi, MD, Principal Investigator — E.O. Ospedali Galliera
Locations (1):
- E.O. Ospedali Galliera, Genova, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the primary publication of the trial will be shared (text, tables, figures, and appendices), after deidentification
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared 3 months following the publication of the article and they will remain available for 36 months.
Access Criteria: the investigators who would like to use the data have to prepare a proposal that should be send to the Principal investigator (andrea.decensi@galliera.it).To gain access, data requestors will need to sign a data access agreement

REFERENCES:
- [Derived] Buttiron Webber T, Provinciali N, Musso M, Ugolini M, Boitano M, Clavarezza M, D'Amico M, Defferrari C, Gozza A, Briata IM, Magnani M, Paciolla F, Menghini N, Marcenaro E, De Palma R, Sacchi N, Innocenti L, Siri G, D'Ecclesiis O, Cevasco I, Gandini S, DeCensi A. Predictors of poor seroconversion and adverse events to SARS-CoV-2 mRNA BNT162b2 vaccine in cancer patients on active treatment. Eur J Cancer. 2021 Dec;159:105-112. doi: 10.1016/j.ejca.2021.09.030. Epub 2021 Oct 11. PMID 34742157